CLINICAL TRIAL: NCT01954836
Title: Short-Term Fasting During Chemotherapy in Patients With Gynecological Cancer- a Randomized Controlled Cross-over Trial
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof.Dr.med Andreas Michalsen, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FIT08/2013
Record Dates: First submitted 2013-09-29; First posted 2013-10-07 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasia; Cancer; Fasting
Keywords: short-term fasting; adjuvant chemotherapy; toxicity; side-effects; ovarial carinoma; breast cancer
MeSH Terms: conditions — Neoplasms; Fasting; Intermittent Fasting; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initial fasting (Experimental): Fasting during chemotherapy of the first half of chemotherapy cycles (1 and 2 of four or 1 to 3 of six cycles)
  Interventions: Behavioral: initial fasting
- Secondary fasting (Active Comparator): Fasting during the second half of chemotherapy cycles (3 and 4 of four cycles or 4 to 6 of six cycles)
  Interventions: Behavioral: Secondary fasting

INTERVENTIONS:
Behavioral: initial fasting — modified fasting with daily caloric intake of <400kcal by juices starting 36 to 48 h before begin of chemotherapy and lasting to 24 h after end of chemotherapy applied in the first half of scheduled 4 or 6 chemotherapy cycles
  Arms: Initial fasting
Behavioral: Secondary fasting — modified fasting with daily caloric intake of <400kcal by juices starting 36 to 48 h before begin of chemotherapy and lasting to 24 h after end of chemotherapy applied in the second half of scheduled 4 or 6 chemotherapy cycles
  Arms: Secondary fasting

SUMMARY:
Hypothesis: Fasting before (48h) and one day after chemotherapy may protect normal cells from the adverse effects of chemotherapy. Design: Within a randomized controlled pilot trial 30 female patients with gynecological cancer (ovarian and breast cancer)and 4-6 scheduled chemotherapies will be randomized to fast 60-72 hours during the first half of chemotherapies or during the second half of chemotherapies and to proceed normocaloric food intake during the other cycles.Sequence of fasting and normocaloric food intake will be randomized. Assessments of adverse effects, quality of life and laboratory values take place 24 and 7 days after each chemotherapy. Statistical analyses compare summarized differences of fasted and non-fasted chemotherapy cycles.

DETAILED DESCRIPTION:
Evidence from experimental animals provides strong support for the concept that caloric restriction (CR) increases resistance to multiple forms of stress. CR decreases plasma levels of growth factors, e.g. insulin-like growth factor-I (IGF-I), thereby diverting energy from growth to maintenance. Accordingly, the currently available information suggests that short-term fasting protects normal cells against the perils of (high dose) chemotherapy. In contrast, cancer cells are not (or less) protected as a result of their self-sufficiency in growth signals. This phenomenon is termed Differential Stress Resistance (DSR). DSR may reduce the severity of adverse effects caused by chemotherapy, without interfering with its anti-tumoral effects. A first case series of 10 cancer patients, suggested that short-term fasting may also protect against the side effects of chemotherapy in humans. This study aims to further evaluate the impact of short-term fasting on tolerance to chemotherapy in humans.Within a randomized controlled pilot trial 30 female patients with gynecological cancer disease (ovarian and breast cancer)in all stages and 4-6 scheduled chemotherapies will be randomized to fast 60-72 hours during half of chemotherapies and to have normocaloric food intake during the other chemotherapies. Fasting is defined as caloric restriction to below 400kcal energy intake/day with free intake of water and tea. Sequences of fasting and normocaloric food intake will be randomized. Assessments of adverse effects, quality of life, fatigue and laboratory values will take place 24 and 7 days after each chemotherapy. Statistical analyses will compare the summarized differences of fasted and non-fasted chemotherapy cycles, that means a total of max. 60-90 chemotherapies with accompanying fasting will be compared to 60-90 non-fasted chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian cancer or breast cancer
* scheduled chemotherapy
* First diagnosis or 1.recurrence

mono

Exclusion Criteria:

* cachexia (BMI < 21kg/m2)
* eating disorder
* renal failure (Crea >2mg/dl)
* enterostoma
* short bowel syndrome
* not assigned to other studies

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Quality of life, modified FACT-O | 24 h and 7 days after chemotherapy cycle

SECONDARY OUTCOMES:
Fatigue | 24 h and 7 days after chemotherapy cycle
Intensity of adverse effects structured criteria Likert scales | 24 h and 7 days after chemotherapy cycles
Laboratory assessments (blood count, liver, renal function) | 24 h and 7 days after chemotherapy cycles

CONTACTS AND LOCATIONS:
Overall Officials: andreas A Michalsen, M.D., Principal Investigator — Charite University
Locations (1):
- Charite University, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauersfeld SP, Kessler CS, Wischnewsky M, Jaensch A, Steckhan N, Stange R, Kunz B, Bruckner B, Sehouli J, Michalsen A. The effects of short-term fasting on quality of life and tolerance to chemotherapy in patients with breast and ovarian cancer: a randomized cross-over pilot study. BMC Cancer. 2018 Apr 27;18(1):476. doi: 10.1186/s12885-018-4353-2. PMID 29699509